CLINICAL TRIAL: NCT02870452
Title: Effectiveness of Two Psychological Interventions for Prevention and Management of Pain, Emotional Regulation and Promotion of Quality of Life in People With Haemophilia: a Randomized Controlled Trial
Brief Title: Effectiveness of Psychological Interventions in Haemophilia
Acronym: PSY_HaEMOPEQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Patrícia Ribeiro Pinto, Post-doctoral fellow, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RCT520101.ID1825
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Haemophilia
Keywords: Haemophilia; RCT; Pain; Hemarthrosis; Hypnosis; Cognitive-Behavioral Therapy; Quality of Life; Distress; Cytokines
MeSH Terms: conditions — Hemophilia A; Pain; Hemarthrosis | interventions — Hypnosis; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis (Experimental): Hypnosis for the prevention and management of pain, emotional regulation and promotion of quality of life in people with Haemophilia
  Interventions: Behavioral: Hypnosis
- Cognitive-Behavioral Therapy (Experimental): Cognitive Behavioral Therapy for the prevention and management of pain, emotional regulation and promotion of quality of life in people with Haemophilia
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Control Group (No Intervention): No psychological intervention - standard Haemophilia care

INTERVENTIONS:
Behavioral: Hypnosis — 4 weekly individual sessions of Hypnosis, conducted by a certified psychologist, with the approximate duration of 90 minutes.
  Arms: Hypnosis
Behavioral: Cognitive-Behavioral Therapy — 4 weekly individual sessions of CBT, conducted by a certified psychologist, with the approximate duration of 90 minutes.
  Arms: Cognitive-Behavioral Therapy

SUMMARY:
The purpose of this study is to evaluate the relative effectiveness of two psychological interventions, cognitive-behavioral therapy (CBT) and hypnosis (Hyp), in preventing and managing pain, regulating emotional state and improving quality of life in Portuguese PWH.

DETAILED DESCRIPTION:
22 (People with Haemophilia) PWH will be included in each group (Hypnosis, CBT and control-no intervention) (total=66). Sample size was calculated using G*Power 3.1.4 and considering the following assumptions: to perform a one-way ANOVA with fixed effects, a large effect size (f =0.4), a significance level (α - type I error) of 0.05 and a statistical power (1-β - type II error) of 0.80.

The patients will be approached by clinicians of the Immunohaemotherapy Department and the psychologists for the explanation of the study, confidentiality and voluntary nature of participation. Patients who agree to participate will be asked to read and sign the Informed Consent document. Afterwards, the first assessment moment will take place in order to get a baseline assessment of each patient (T0: pre-test). Subsequently, the blind randomization to one of the 3 conditions will occur and the 4 individual intervention sessions will be scheduled, occurring in a weekly basis (90 minutes per session).

The post-test assessment (T1) takes place one week after the last intervention session (in the 5th week), and the follow-up assessments (T2, T3 and T4) will occur subsequently at 3 months, 6 months and one year post-intervention.

A physiological assessment will be performed at T1, T2 and T4. This will be performed through the collection of blood samples in order to achieve a systemic evaluation of pro-inflammatory and anti-inflammatory cytokines. A CBC (Complete Blood Count) with White Blood Count and C Reactive Protein (CRP) analysis will also be performed. Upon arrival at the Immunohaemotherapy Department (between 9:30 am and 1:30 pm), patients will undergo sample blood collection and EDTA-samples will be transported immediately to the lab.

In the lab, blood samples are centrifuged 15 minutes at 3.000 rpm, and plasma aliquoted and stored in a freezer at -80 ºC, until further analysis. Plasma levels of cytokines (IL-6, IL-1β, TNF-α, IL-10) are assayed in duplicate using ultra-sensitive multiplex human ELISA kits (Life Technologies®).

Functional Assessment of the joints will be performed through the Gilbert (based on clinical evaluation) and Pettersson Scores (based on X-ray and ultrasonography).

All study procedures will comply with the applicable ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Mild pr severe Haemophilia A or B
* Age of 18 or older
* Ability to write and read

Exclusion Criteria:

* Other comorbid life threatening diseases, such as cancer
* Neurological or psychiatric deficits
* Acquired Haemophilia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity at 1 week as assessed by Numeric Rating Scale (NRS) | 1 week post-intervention
Pain intensity at 3 months as assessed by NRS | 3 months post-intervention
Pain intensity at 6 months as assessed by NRS | 6 months post-intervention
Pain intensity at 12 months as assessed by NRS | 12 months post-intervention

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQOL) at 1 week as assessed by A36Hemofilia-Qol | 1 week
HRQOL at 3 months as assessed by A36Hemofilia-Qol | 3 months
HRQOL at 6 months as assessed by A36Hemofilia-Qol | 6 months
HRQOL at 12 months as assessed by A36Hemofilia-Qol | 12 months
Haemophilia related functional limitations at 1 week as assessed by Haemophilia Activities List (HAL) | 1 week
Haemophilia related functional limitations at 3 months as assessed by HAL | 3 months
Haemophilia related functional limitations at 6 months as assessed by HAL | 6 months
Haemophilia related functional limitations at 12 months as assessed by HAL | 12 months
Anxiety at 1 week as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-Anxiety Short Form v1.0 | 1 week
Anxiety at 3 months as assessed by PROMIS-Anxiety Short Form v1.0 | 3 months
Anxiety at 6 months as assessed by PROMIS-Anxiety Short Form v1.0 | 6 months
Anxiety at 12 months as assessed by PROMIS-Anxiety Short Form v1.0 | 12 months
Depression at 1 week as assessed by PROMIS-Depression Short Form v1.0 | 1 week
Depression at 3 months as assessed by PROMIS-Depression Short Form v1.0 | 3 months
Depression at 6 months as assessed by PROMIS-Depression Short Form v1.0 | 6 months
Depression at 12 months as assessed by PROMIS-Depression Short Form v1.0 | 12 months
Pain Catastrophizing at 1 week as assessed by Coping Strategies Questionnaire (CSQ) Catastrophizing Subscale | 1 week
Pain Catastrophizing at 3 months as assessed by CSQ Catastrophizing Subscale | 3 months
Pain Catastrophizing at 6 months as assessed by CSQ Catastrophizing Subscale | 6 months
Pain Catastrophizing at 12 months as assessed by CSQ Catastrophizing Subscale | 12 months
Illness Perception (Personal Control) at 1 week as assessed by Revised Illness Perception Questionnaire (IPQ-R) | 1 week
Illness Perception (Emotional Representation) at 1 week as assessed by IPQ-R | 1 week
Illness Perception (Personal Control) at 3 months as assessed by IPQ-R | 3 months
Illness Perception (Emotional Representation) at 3 months as assessed by IPQ-R | 3 months
Illness Perception (Personal Control) at 6 months as assessed by IPQ-R | 6 months
Illness Perception (Emotional Representation) at 6 months as assessed by IPQ-R | 6 months
Illness Perception (Personal Control) at 12 months as assessed by IPQ-R | 12 months
Illness Perception (Emotional Representation) at 12 months as assessed by IPQ-R | 12 months
Number of joint bleeds in the previous month, at 1 week | 1 week
Number of joint bleeds in the previous month, at 3 months | 3 months
Number of joint bleeds in the previous month, at 6 months | 6 months
Number of joint bleeds in the previous month, at 12 months | 12 months
Analgesic intake in the previous month, at 1 week | 1 week
Analgesic intake in the previous month, at 3 months | 3 months
Analgesic intake in the previous month, at 6 months | 6 months
Analgesic intake in the previous month, at 12 months | 12 months
Replacement factor (VIII/IX) consumption in the previous month, at 1week | 1 week
Replacement factor (VIII/IX) consumption in the previous month, at 3 months | 3 months
Replacement factor (VIII/IX) consumption in the previous month, at 6 months | 6 months
Replacement factor (VIII/IX) consumption in the previous month, at 12 months | 12 months
Pettersson Score at 3 months | 3 months
  Radiologic classification of PWH joint status
Pettersson Score at 12 months | 12 months
  Radiologic classification of PWH joint status
Gilbert Score at 3 months | 3 months
  Joint health evaluation, in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in hemophilia - knees, ankles, elbows
Gilbert Score at 12 months | 12 months
  Joint health evaluation, in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in hemophilia - knees, ankles, elbows
IL-6 Cytokine at 3 months | 3 months
IL-6 Cytokine at 12 months | 12 months
IL-1β Cytokine at 6 months | 6 months
IL-1β Cytokine at 12 months | 12 months
IL-10 Cytokine at 6 months | 6 months
IL-10 Cytokine at 12 months | 12 months
TNF-α Cytokine at 6 months | 6 months
TNF-α Cytokine at 12 months | 12 months
C Reactive Protein at 6 months | 6 months
C Reactive Protein at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia R Pinto, PhD, Principal Investigator — Life and Health Sciences Research Institute
Locations (1):
- Life and Health Sciences Research Institute, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinto PR, Paredes AC, Costa P, Carvalho M, Lopes M, Fernandes S, Pedras S, Almeida A. Effectiveness of two psychological interventions for pain management, emotional regulation and promotion of quality of life among adult Portuguese men with haemophilia (PSY-HaEMOPEQ): study protocol for a single-centre prospective randomised controlled trial. BMJ Open. 2017 Sep 3;7(9):e016973. doi: 10.1136/bmjopen-2017-016973. PMID 28871021